CLINICAL TRIAL: NCT03947775
Title: A Multicenter, Randomized Controlled Trial of the Efficacy, Safety and Immunogenicity of HPV Vaccination in Preventing Recurrence of HSIL in HIV-positive MSM
Brief Title: HPV-SAVE_Merck_Sub-Study for Preventing Recurrence of HSIL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Irving Salit, Immunodeficiency Clinic, Toronto General Hospital, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 53205
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Anal Intraepithelial Neoplasia; Anal Cancer; Human Papilloma Virus
Keywords: Men who have sex with men; Human immunodeficiency virus; Human papillomavirus; Vaccine; Gardasil; Anal Intraepithelial Neoplasia; Anal Cancer; 9-valent
MeSH Terms: conditions — Anus Neoplasms; Homosexuality; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: This will be a randomized, open-label multicentre clinical trial consisting of two arms (immediate versus delayed vaccination) assessing the efficacy, safety and immunogenicity of the 9-valent recombinant HPV vaccine in HIV-positive males 18 years of age and older. The delayed arm will receive Gardasil-9 12 months after the immediate arm. Similarly, appropriate follow-ups and testing in the delayed arm will occur 12 months after the immediate arm.
  Participants for the proposed study will be recruited from Canadian centres in Toronto, and Vancouver through ongoing projects making up our HPV-SAVE team grant. Other study sites may be added as the study progresses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Vaccination (Experimental): Administration of dose #1 of 9-valent HPV vaccination will be given at baseline visit, dose #2 at month 2, and dose #3 at month 6.
  Interventions: Drug: 9-valent HPV vaccination
- Delayed Vaccination (Active Comparator): Administration of dose #1 of 9-valent HPV vaccination will be given at month 12, dose #2 at month 14, and dose #3 at month 18.
  Interventions: Drug: 9-valent HPV vaccination

INTERVENTIONS:
Drug: 9-valent HPV vaccination — Gardasil-9 is a novel, 9-valent HPV recombinant vaccine, which expands the coverage of oncogenic HPV types, with the addition of HPV types 31, 33, 45, 52, and 58 to the existing quadrivalent vaccine types. The addition of these five oncogenic types is estimated to improve cancer coverage to 90% (versus 70% for the quadrivalent vaccine) [38]. With its expanded coverage of oncogenic HPV types, its proven efficacy in primary prevention and its potential role in mitigating HGAIN recurrences.
  Other Names: Gardasil-9

SUMMARY:
Human papillomavirus (HPV) is the most common sexually transmitted infection (STI) worldwide. Infection by certain high-risk oncogenic types of HPV (HR-HPV) is the major cause of several cancers in men, notably squamous cell carcinoma (SCC) of the anal canal. Rates of anal infection with these HR-HPV strains, and the resultant high-grade anal dysplasia and anal cancer are much higher in men who have sex with men (MSM) than in the general population. Co-infection with human immunodeficiency virus (HIV) further amplifies this burden, making the rates of anal SCC in HIV-positive MSM higher than the historic rates of cervical cancer prior to the adoption of routine cervical cytology screening. Despite these alarming statistics, there are no established protocols for optimal screening and treatment of anal HPV and cancer precursors, nor has there been any widespread rollout of organized screening programs anywhere in Canada. Further, not only does HPV directly cause significant disease in these men, but there is growing epidemiologic evidence that HPV infection may enhance sexual transmission of HIV. These significant knowledge gaps translate into fundamental deficiencies in care for HIV-positive MSM.

The HPV Screening and Vaccine Evaluation in MSM (HPV-SAVE) study team was funded by the Canadian Institutes of Health Research (CIHR) via its Boys' and Men's Health Team Grant Competition. It aims to recruit a large group of MSM from various Ontario and Vancouver clinics, in order to carry out a number of different studies. The HPV-SAVE team brings together community and internationally-recognized experts in HPV and HIV disease and mucosal immunology, to better define the optimal approaches for primary and secondary prevention and treatment of HPV-associated anal disease among HIV-positive MSM, and to explore biological mechanistic evidence regarding the potential role of HPV as a co-factor for HIV transmission. This will yield critical information which can lead to improvement in the health of MSM, and will provide a foundation on which to build large-scale screening and treatment trials on a national level. A key part of this research program involves an analysis of the potential role played by the HPV vaccine in the overall management of HIV-positive MSM.

Planned vaccine-related projects include:

* A mixed-methods analysis of the knowledge, attitudes, and acceptability of HPV vaccination amongst HIV-positive MSM, through quantitative (e.g. cross-sectional survey) and qualitative (e.g. in-depth interviews) means.
* A comprehensive assessment of the 9-valent HPV vaccine in HIV-positive MSM, including safety and immunogenicity, as well as its potential role in secondary prevention of high-grade anal dysplasia. This is the study on which the current proposal is based.

DETAILED DESCRIPTION:
Advances in the treatment of HIV-infected individuals with the advent of the combination antiretroviral therapy (cART) era has led to dramatic reductions in mortality and morbidity. These dramatic strides in survival within HIV-positive populations have led to a focus on longer-term morbidities in these individuals, including malignancies. Indeed, an increase in a variety of malignancies in HIV-infected individuals has been noted in the cART era. Amongst these are cancers associated with HPV, responsible for the vast majority of cervical cancers (itself a well-established acquired immune deficiency syndrome (AIDS)-defining illness), and 40-90% of anal, vulvar, vaginal, penile, and oropharyngeal cancers. More specifically, a recent meta-analysis indicates that the overall prevalence of HPV in anal carcinoma is approximately 84%, with HPV type 16 being isolated in 73% of all cases, making it the most prevalent type implicated in anal carcinoma.

Though infrequent at a rate of one per 100 000, squamous cell anal carcinoma is on the rise in the general population. It occurs at significantly higher rates in HIV-positive men - particularly among MSM - with an estimated rate of 60 to 160 per 100 000. A recent study of thirteen North American AIDS Cohort Collaboration on Research and Design (NA-ACCORD) with over 34,000 HIV-infected patients, found that anal cancer rates were highest in HIV-infected MSM, with a rate of 131 per 100,000 person years. In fact, rates of anal cancer among HIV-infected MSM are comparable to rates of cervical cancer in women prior to the adoption of routine screening for cervical dysplasia. In addition to its etiologic association with HPV, anal cancer shares many similarities with cervical cancer. Both are squamous cell cancers occurring at the squamo-columnar junction, and both likely arise from histologically-similar, dysplastic precursor lesions. It is postulated that a critical step in anal cancer carcinogenesis is the establishment of persistent infection (conventionally defined as greater than six or twelve months) with oncogenic HPV in the anal canal. Though the majority of HPV infections are considered transient and will eventually clear even in HIV-positive individuals, HIV-positive individuals have higher rates of persistent infection, especially with oncogenic HPV types.

Of the greater than 170 HPV types, over 30 favour the anogenital area, and on the basis of epidemiologic and phylogenetic data, these have been classified by the International Agency for Research on Cancer (IARC).

The vast majority of anal cancers (as well as cervical cancers) are caused by two high-risk HPV types: HPV type 16 and HPV type 18, felt to be responsible for 66% and 5% of anal cancers, respectively. However, a recent study from France examining the distribution of HPV types in cases of anal cancer found even more dramatic results: HPV was found in 96.7% of all cases, with HPV-16 being the most prevalent type (75%), with other high risk types (HPV-18, -52, -33, and -51) found in 4% to 6% of cases. Further, HPV-16 and -18 - either alone or in combination - were found in over 78% of cases. HPV lesions caused by low-risk types include condylomata (or commonly known as 'genital warts'), of which 90% are caused by HPV types 6 and 11.

Prevention strategies for anal cancers have emerged that are analogous to strategies used in cervical cancer screening, that rely on a combination of cytology (Papanicolaou, or Pap smear) and high-resolution anoscopy (HRA; analogous to colposcopy), both of which screen for high-grade anal intraepithelial neoplasia (HGAIN; typically graded as anal intraepithelial neoplasia (AIN) AIN-2 or -3). Despite the clear evidence indicating the benefit of screening and treatment procedures in cervical cancer screening, no large rigorous studies have been performed to assess the performance of such strategies in anal cancer screening in either men or women.

In addition to the scant literature on the efficacy of screening programs for anal cancer and HPV in all men - but particularly those who are HIV-positive - there remains an even greater paucity of data on issues surrounding primary prevention of HPV. The HPV quadrivalent recombinant vaccine, or Gardasil®, protects against HPV types 6 and 11, which are the most common types implicated in condylomata acuminata (anogenital warts), as well as the most common oncogenic strains, types 16 and 18. The use of this vaccine has been shown to prevent persistent cervical HPV infection caused by vaccine types in women, as well as preventing nearly all high grade genital lesions in women - the latter of which are considered precursor lesions to invasive cancers. Additionally, a retrospective pooled analysis of two large efficacy trials of quadrivalent HPV vaccine has also demonstrated a treatment effect from HPV vaccine in preventing recurrences of previously treated high grade cervical disease.

Few studies have been done on the use of the quadrivalent HPV vaccine in men; there has only been one study examining the use of the HPV vaccine in HIV-positive men, and this study found the vaccine to be safe and immunogenic. Overall, these studies have shown promise, demonstrating a reduction in vaccine-type genital lesions in young men who were vaccinated versus those receiving placebo, evidence of protection against HGAIN in MSM, and a 50% reduction rate in HGAIN recurrence in MSM previously treated for dysplastic lesions. This latter study lays the foundation of the currently proposed study. However, the role of the HPV vaccine in secondary prevention of HGAIN has not been examined in a systematic, prospective way. Given the unacceptably high rates of HGAIN recurrence in those having undergone ablative therapy (from 62% to 91% within two years in HIV-positive MSM), exploring this potentially novel benefit of the HPV vaccine is certainly warranted and could potentially change the way clinicians address HPV-related disease in this high-risk group.

Until recently there existed no standard recommendation for the use of HPV vaccinations in males, regardless of HIV serostatus; however, these studies have prompted the Centres for Disease Control and Prevention's (CDC) Advisory Committee on Immunization Practices (ACIP) to recommend that boys be routinely vaccinated for HPV beginning at age 11 or 12. Canada's National Advisory Committee on Immunizations (NACI) went further, recommending vaccination in all males between 9 and 26 years of age, as well as any MSM 9 years of age or older.

Gardasil-9 is a novel, 9-valent HPV recombinant vaccine, which expands the coverage of oncogenic HPV types, with the addition of HPV types 31, 33, 45, 52, and 58 to the existing quadrivalent vaccine types. The addition of these five oncogenic types is estimated to improve cancer coverage to 90% (versus 70% for the quadrivalent vaccine). With its expanded coverage of oncogenic HPV types, its proven efficacy in primary prevention and its potential role in mitigating HGAIN recurrences - all coupled with the disproportionate burden of HPV-related anal cancers borne by HIV-positive MSM - it is critical that its use be comprehensively assessed in this very high risk population

ELIGIBILITY:
Subject Inclusion Criteria

1. Males, aged ≥ 18 years at baseline;
2. Physician or laboratory documentation of HIV-1 infection (enzyme-linked immunosorbent assay [ELISA] and Western Blot);
3. AIN-2 or -3 found on biopsy of anal canal lesion(s), and willingness of the subject to undergo ablative therapy which is standard of care in most screening clinics;
4. History of any sexual activity with men, or both men and women, where sexual activity is defined as oral, vaginal, or anal intercourse;
5. For those on cART, the participant must be on a stable regimen (i.e. virologically suppressed with HIV-1 ribonucleic acid (RNA) below the assay's limit of detection for minimum six months). This will minimize confounding from dramatic shifts in viral load and/or cluster of differentiation 4 (CD4) count;
6. For those individuals that are not on cART, there must be no immediate plans to initiate cART in the next six months. There will be no lower limit cut-off for CD4 count;
7. An ability to give informed consent;
8. An ability to attend clinic for all study visits.

Subject Exclusion Criteria

1. Known hypersensitivity to any component of the HPV vaccine (e.g. Saccharomyces cerevisiae yeast, Amorphous Aluminium Hydroxyphosphate Sulfate adjuvant);
2. Current or prior history of cancer of the anogenital regions (e.g. penile, anal, or rectal) or of the oropharyngeal area (e.g. oral cavity, upper airway).
3. Previous HPV immunization.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — History of any sexual activity with men, or both men and women, where sexual activity is defined as oral, vaginal, or anal intercourse.
Enrollment: 228 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants in each arm with biopsy-proven HGAIN (AIN-2/3). | 24 months, following successful treatment of HGAIN
  Secondary Prevention. "Successful treatment" refers to a biopsy-proven HGAIN lesion treated with ablative therapy electrocautery (EC) with repeat biopsy of the same lesion 2-3 months thereafter demonstrating no further evidence of HGAIN (meaning that the follow-up biopsy is either AIN-1 or normal).

SECONDARY OUTCOMES:
The geometric mean titres (GMT) of antibody to each vaccine type above a pre-specified, validated cut-off. F | 24 months, following successful treatment of HGAIN
  Immunogenicity. or this measure, immunogenicity will be measured as the proportion of participants with GMT of antibody to each vaccine type above a pre-specified, validated cut-off, using a Luminex-based immunoassay [40-42]. Currently, these values for the HPV types present in the 9-valent vaccine are: HPV-6, 30 milli-Merck units/ml (mMU/mL); HPV-11, 16 mMU/mL; HPV-16, 20 mMU/mL; HPV-18, 24 mMU/mL; HPV-31, 10 mMU/mL; HPV-33, 8 mMU/mL; HPV-45, 8 mMU/mL; HPV-52, 8 mMU/mL; and HPV-58, 8 mMU/mL .

OTHER OUTCOMES:
Change in anal carriage of vaccine HPV types. Repeated detection of anal HPV will indicate the duration of carriage. This will be compared between the early and delayed vaccine groups. | 24 months
  Immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Irving Salit, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (4):
- Canada (4):
  - BC Centre for Disease Control, Vancouver, British Columbia
  - University of British Columbia, Vancouver, British Columbia
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Background] Palella FJ Jr, Delaney KM, Moorman AC, Loveless MO, Fuhrer J, Satten GA, Aschman DJ, Holmberg SD. Declining morbidity and mortality among patients with advanced human immunodeficiency virus infection. HIV Outpatient Study Investigators. N Engl J Med. 1998 Mar 26;338(13):853-60. doi: 10.1056/NEJM199803263381301. PMID 9516219
- [Background] Hammer SM, Eron JJ Jr, Reiss P, Schooley RT, Thompson MA, Walmsley S, Cahn P, Fischl MA, Gatell JM, Hirsch MS, Jacobsen DM, Montaner JS, Richman DD, Yeni PG, Volberding PA; International AIDS Society-USA. Antiretroviral treatment of adult HIV infection: 2008 recommendations of the International AIDS Society-USA panel. JAMA. 2008 Aug 6;300(5):555-70. doi: 10.1001/jama.300.5.555. PMID 18677028
- [Background] Chiao EY, Krown SE, Stier EA, Schrag D. A population-based analysis of temporal trends in the incidence of squamous anal canal cancer in relation to the HIV epidemic. J Acquir Immune Defic Syndr. 2005 Dec 1;40(4):451-5. doi: 10.1097/01.qai.0000159669.80207.12. PMID 16280701
- [Background] Swedish KA, Factor SH, Goldstone SE. Prevention of recurrent high-grade anal neoplasia with quadrivalent human papillomavirus vaccination of men who have sex with men: a nonconcurrent cohort study. Clin Infect Dis. 2012 Apr;54(7):891-8. doi: 10.1093/cid/cir1036. Epub 2012 Jan 30. PMID 22291111
- [Background] Joura EA, Garland SM, Paavonen J, Ferris DG, Perez G, Ault KA, Huh WK, Sings HL, James MK, Haupt RM; FUTURE I and II Study Group. Effect of the human papillomavirus (HPV) quadrivalent vaccine in a subgroup of women with cervical and vulvar disease: retrospective pooled analysis of trial data. BMJ. 2012 Mar 27;344:e1401. doi: 10.1136/bmj.e1401. PMID 22454089